CLINICAL TRIAL: NCT04612517
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Subcutaneous Doses of ZP7570 in Healthy Subjects
Brief Title: A Multiple Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP7570
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZP7570-18145; 2019-001129-29 (EudraCT Number)
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, single ascending dose trial in healthy subjects, randomized to ZP7570 or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP7570 (Experimental): Four ascending doses of ZP7570
  Interventions: Drug: ZP7570
- Placebo (Placebo Comparator): Corresponding volume of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP7570 — Each subject will be randomly allocated to multiple doses of ZP7570 at one of four dose levels in each cohort.
  Other Names: Dual GLP-1R/GLP-2R agonist
  Arms: ZP7570
Drug: Placebo — Placebo; corresponding volume
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multiple ascending dose trial in healthy subjects, randomised to ZP7570 or placebo within each cohort

DETAILED DESCRIPTION:
Forty subjects are planned to be studied in four cohorts in this multiple ascending dose trial. Ten subjects will be allocated to four dose levels. Intermediate dose levels may be applied. A sentinel dosing approach (sequential dosing) will be applied. The entire observation period comprises 51 days starting with a 96 hours in-house stay after the first dose injection, where discharge is planned for Day 5, followed by one outpatient visit. For the second and the third injection dose a 36 hours in-house stay is planned. After the fourth dose injection there is also a 96 hour in-house stay where discharge is planned for Day 26, followed by five outpatient visits and an End of Trial Visit on Day 51. A blinded evaluation of each cohort will be performed by a Trial Safety Group to determine whether the trial will progress to the next planned dose level based on the stopping rules specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the subject.
* Healthy male or female subject (only women not of childbearing potential) aged between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 28.0 kg/m2, both inclusive
* A body weight of at least 60 kg.
* Heart rate after 5 minutes rest in supine position inside the range of 50-90 beats/min at screening

Exclusion Criteria:

* Any history of a disorder which in the investigator's opinion might jeopardize subjects safety, evaluation of results or compliance with the protocol.
* History of gallbladder disease or cholecystectomy.
* History of pancreatitis
* History of major depressive disorder or a Patient Health Questionnaire (PHQ-9) > 9 completed at screening, or a history of other severe psychiatric disorders (e.g. schizophrenia or bipolar disorder).
* Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to screening.
* Family history of multiple endocrinological neoplasia type 2 (MEN2) or medullary thyroid carcinoma (MTC).
* Clinically significant abnormal standard 12-lead ECG after 5 min resting in supine position at screening, including a QTcF > 450 ms (males) or QTcF > 470 ms (females), PR ≥ 220 ms and QRS ≥ 110 ms.
* History of severe hypersensitivity to medicines or foods or history of severe medicinal/food induced anaphylactic reaction .
* Any clinically significant abnormal hematology, biochemistry, or urinalysis screening tests, as judged by the investigator.
* TSH values outside of normal reference ranges of safety laboratory
* Estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73 m2, as defined by - Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
* Known or suspected hypersensitivity to IMP(s) or related products.
* Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension).
* Symptoms of arterial hypotension
* Women of childbearing potential
* Men with non-pregnant partner(s) of childbearing potential not willing to use male contraception (condom) in addition to a highly effective contraceptive method until 28 days after dosing
* Men with pregnant partner not willing to use male contraception (condom) until 28 days after dosing, in order to avoid exposure of the embryo/fetus to seminal fluid.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability - Incidence of treatment emergent adverse events as assessed by type and severity | From time 0 to 51 days after first dosing (29 days after fourth dosing) ]
  The incidence, type and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics - Area under the plasma concentration-time curve - through | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  AUCτ, Area under the plasma concentration-time curve from zero to through concentration.
Pharmacokinetics - Area under the plasma concentration-time curve - infinity | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  AUCinf, Area under the plasma concentration-time curve from zero to infinity concentration.
Pharmacokinetics - Area under the plasma concentration-time curve - last | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  AUClast, Area under the plasma concentration-time curve-from zero to last concentration.
Pharmacokinetics - Maximum plasma concentration - Cmax | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Cmax, Measured maximum plasma drug concentration after dosing
Pharmacokinetics - Time to maximum plasma concentration - Tmax | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Tmax, Sampling time until reaching Cmax after dosing
Pharmacokinetics - Elimination rate constant - λz | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  λz, Elimination rate constant
Pharmacokinetics - Half-life - t½ | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  t½, Half-life of ZP7570
Pharmacokinetics - Volume of distribution - Vz/f | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Vz/f, Apparent volume of distribution of ZP7570 during terminal phase
Pharmacokinetics - Body clearance - CL/f | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  CL/f, Apparent total body clearance
Pharmacokinetics - Mean residence time - MRT | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  MRT, Mean residence time
Pharmacodynamics - Acetaminophen concentration-time curves | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the the forth dose
  Acetaminophen concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum acetaminophen concentration - Cmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the the forth dose
  Cmax, maximum acetaminophen concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum acetaminophen concentration - Tmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum acetaminophen concentration following ingestion of mixed meal test and acetaminophene
Pharmacodynamics - Area under the concentration-time curve - AUCacetaminohen,0-60min | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the the forth dose
  AUCacetaminohen,0-60min, area under the acetaminophen concentration-time curve from 0 to 60 min post-ingestion
Pharmacodynamics - Area under the concentration-time curve - AUCacetaminohen,0-240min | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCacetaminohen,0-240min, area under the acetaminophen concentration -time curve from 0 to 240 min post-ingestion
Pharmacodynamics - Plasma glucose concentration-time curves | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the the forth dose
  Plasma glucose concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum plasma glucose concentration - Cmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the the forth dose
  Cmax, Maximum plasma glucose concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum plasma glucose concentration - Tmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum plasma glucose concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Area under the concentration-time curve - AUCplasma glucose,0-60min | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCplasma glucose,0-60min, area under the plasma glucose concentration-time curve from 0 to 60 min post-ingestion
Pharmacodynamics - Area under the concentration-time curve - AUCplasma glucose,0-240min | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCplasma glucose,0-240min, area under the acetaminophen concentration -time curve from 0 to 240 min post-ingestion
Pharmacodynamics - Insulin concentration-time curves | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Insulin concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum insulin concentration - Cmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Cmax, Maximum insulin concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum insulin concentration - Tmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum insulin concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Area under the concentration-time curve - AUCinsulin,0-60min | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCinsulin,0-60min, area under the insulin concentration-time curve from 0 to 60 min post-ingestion
Pharmacodynamics - Area under the concentration-time curve - AUCinsulin, 0-240min | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCinsulin,0-240min, area under the insulin concentration-time curve from 0 to 240 min post-ingestion
Pharmacodynamics - Glucagon concentration-time curves (optional) | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Glucagon concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum glucagon concentration - Cmax (optional) | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Cmax, Maximum glucagon concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum glucagon concentration - Tmax (optional) | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum glucagon concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Area under the concentration-time curve - AUCglucagon,0-60min (optional) | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCglucagon,0-60min, area under the glucagon concentration-time curve from 0 to 60 min post-ingestion
Pharmacodynamics - Area under the concentration-time curve - AUCglucagon, 0-240min (optional) | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCglucagon,0-240min, area under the glucagon concentration-time curve from 0 to 240 min post-ingestion
Pharmacodynamics - Free fatty acids concentration-time curves | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Free fatty acids concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum free fatty acids concentration - Cmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Cmax, Maximum free fatty acids concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum free fatty acids concentration - Tmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum free fatty acids concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Area under the concentration-time curve - AUCfree fatty acids, 0-60min | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCfree fatty acids,0-60min, area under the free fatty acids concentration-time curve
Pharmacodynamics - Area under the concentration-time curve - AUCfree fatty acids, 0-240min | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCfree fatty acids,0-240min, area under the free fatty acids concentration-time curve
Pharmacodynamics - Triglycerides concentration-time curves | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Triglycerides concentration-time curves following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Maximum triglycerides concentration - Cmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Cmax, Maximum triglycerides concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Time to maximum triglycerides concentration - Tmax | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  Tmax, Time to maximum triglycerides concentration following ingestion of mixed meal test and acetaminophen
Pharmacodynamics - Area under the concentration-time curve - AUCtriglycerides, 0-60min | From time 0 to 60 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCtriglycerides,0-60min, area under the triglycerides concentration-time
Pharmacodynamics - Area under the concentration-time curve - AUCtriglycerides,0-240min | From time 0 to 240 minutes at baseline, 24 hours after a single dose and 24 hours after the forth dose
  AUCtriglycerides,0-240min, area under the triglycerides concentration-time curve
Anti-ZP7570 antibodies - Incidence and titres | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Overall anti-ZP7570 antibody incidence and titers. Incidence of anti-ZP7570 antibodies cross-reacting with endogenous GLP-1 or GLP-2.
Safety Lab - Haematological values vs. reference ranges and baseline | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Abnormal values or changes in haematology.
Safety Lab - Clinical chemistry values vs. reference ranges and baseline | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Abnormal values or changes in chemical chemistry
Safety Lab - Urinalysis values vs. reference ranges and baseline | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Abnormal values or changes in urinalysis
Safety - Vital signs: blood pressure | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Changes in diastolic and systolic blood pressure (in mmHg)
Safety - Vital signs: pulse | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Changes in pulse (beats per minute)
Safety - Physical Examination | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Changes in physical examination of the body. Outcome will be measured as 'normal' or 'abnormal', if abnormal as 'not clinically significant' or 'clinically significant'.
Safety - ECG | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Changes or abnormalities in ECG parameters (in ms): Heart rate, PR, QRS, QT, QTcF
Safety - Injection site reactions | From time 0 to 51 days after first dosing (29 days after fourth dosing)
  Occurrence of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany